CLINICAL TRIAL: NCT03121586
Title: A 52-Week, Open-Label, Extension Study of Pimavanserin for the Adjunctive Treatment of Schizophrenia
Brief Title: Extension Study of Pimavanserin for the Adjunctive Treatment of Schizophrenia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACP-103-035; 2016-003435-38 (EudraCT Number)
Record Dates: First submitted 2017-04-13; First posted 2017-04-20 (Actual); Results first posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — pimavanserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Drug - Pimavanserin (Experimental): Pimavanserin 34 mg, 20 mg, or 10 mg, + background antipsychotic, taken once daily by mouth
  Interventions: Drug: Pimavanserin

INTERVENTIONS:
Drug: Pimavanserin — Pimavanserin 10 mg, tablet, taken as one 10 mg tablets, once daily by mouth, OR Pimavanserin 20 mg, tablet, taken as two 10 mg tablets, once daily by mouth, OR Pimavanserin 34 mg, tablet, taken as two 17 mg tablets, once daily by mouth

SUMMARY:
To evaluate the long-term safety and tolerability of pimavanserin after 52 weeks of adjunctive treatment in subjects with schizophrenia

ELIGIBILITY:
Inclusion Criteria:

1. Patient is able to understand and provide signed informed consent
2. Has a caregiver or some other identified responsible person (e.g., family member, social worker, caseworker, or nurse) considered reliable by the Investigator in providing support to the subject to help ensure compliance with study treatment, study visits, and protocol procedures and who is also able to provide input helpful for completing study rating scale
3. Is completing the Week 6 visit in Study ACP-103-034 or the Week 26 visit in Study ACP-103-038 or 064 while continuing to take his/her assigned dose of blinded study drug and may, in the Investigator's opinion, benefit from continued adjunctive treatment with pimavanserin to a antipsychotic
4. If the subject is female, she must not be pregnant or breastfeeding. She must also be of non-childbearing potential (defined as either surgically sterilized or at least 1 year postmenopausal) or must agree to use two clinically acceptable methods of contraception
5. The main background antipsychotic with which the subject is being treated must continue to be on one of the antipsychotics listed below:

   * Aripiprazole
   * Aripiprazole long-acting injectables:

     * Abilify Maintena®
     * Aristada®
   * Asenapine
   * Risperidone
   * Risperidone long-acting injection
   * Olanzapine
   * Paliperidone extended release (ER) (≤9 mg)
   * Paliperidone palmitate

     * Invega Sustenna® (≤156 mg)
     * Invega Trinza® (≤546 mg)
     * Trevicta® (≤350 mg)
     * Xeplion® (≤100 mg)
   * Lurasidone
   * Cariprazine
   * Brexpiprazole
   * Asenapine

Exclusion Criteria:

1. Patient is judged by the Investigator or the Medical Monitor to be inappropriate for the study (e.g., significantly noncompliant in Studies ACP-103-034, -038, or -064)
2. A urine drug screen (UDS) result at Baseline that indicates the presence of any tested prohibited substance of potential abuse

   1. Subjects from Studies 034 and 038 with a result indicating the presence of marijuana are permitted, if allowed by medical regulations, if they agree to abstain from marijuana use during the study and the medical monitor approves the subject's participation
   2. Subjects from Study 064 with a result indicating the presence of marijuana are not permitted in the study
3. Is taking a medication or drug or other substance that is prohibited according to this protocol
4. Known family or personal history or symptoms of long QT syndrome or risk factors for torsade de pointes and/or sudden death, including symptomatic bradycardia, hypokalemia or hypomagnesemia, and the presence of congenital prolongation of the QT interval
5. Patient has current evidence of a serious and/or unstable psychiatric, neurologic, cardiovascular, respiratory, gastrointestinal, renal, hepatic, hematologic, or other medical disorder, including cancer or malignancies, which would affect the patient's ability to participate in the study.

Patients will be evaluated at screening to ensure that all criteria for study participation are met. Patients may be excluded from the study based on these assessments (and specifically if it is determined that their baseline health and psychiatric condition do not meet all pre-specified entry criteria).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 995 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (161):
- United States (32):
  - 171-Alea Research Institute, Phoenix, Arizona
  - 156-Woodland International Research Group, LLC, Little Rock, Arkansas
  - 111-Woodland Research Northwest, LLC, Rogers, Arkansas
  - 167-CITrials - Bellflower, Bellflower, California
  - 105-ProScience Research Group, Culver City, California
  - 123-Synergy San Diego, Lemon Grove, California
  - 164-Artemis Institute for Clinical Research, San Diego, California
  - 165-CITrials, Santa Ana, California
  - 108-Collaborative Nueroscience Network, LLC, Torrance, California
  - 125-Galiz Research, Hialeah, Florida
  - 137-Innovative Clinical Research, Inc., Lauderhill, Florida
  - 146-Premier Clinical Research Institute, Inc., Miami, Florida
  - 162-Synexus Clinical Research, Inc., Atlanta, Georgia
  - 168-Atlanta Center for Medical Research, Atlanta, Georgia
  - 102-Northwest Behavioral Research Center, Marietta, Georgia
  - 114-Northwestern University, Chicago, Illinois
  - 101-American Medical Research, Chicago, Illinois
  - 130-Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - 118-Lake Charles Clinical Trials, Lake Charles, Louisiana
  - 124-Altea Research Institute, Las Vegas, Nevada
  - 141-Hassman Research Institute, Berlin, New Jersey
  - 153-Albuquerque Neuroscience Inc., Albuquerque, New Mexico
  - 104-Neurobehavioral Research, Inc., Cedarhurst, New York
  - 140-Synexus Clinical Research, Inc - 140, Jamaica, New York
  - 128-Finger Lakes Clinical Research, Rochester, New York
  - 106-New Hope Clinical Research, Charlotte, North Carolina
  - 145-Carolina Behavioral Care, Durham, North Carolina
  - 110-Cutting Edge Research Group, Oklahoma City, Oklahoma
  - 170-Suburban Research Associates, Downingtown, Pennsylvania
  - 127-University Hills Clinical Research, Irving, Texas
  - 103-Pillar Clinical Research, LLC, Richardson, Texas
  - 115-Psychiatric and Behavioral Solutions LLC, Salt Lake City, Utah
- Argentina (11):
  - 610-Clinica Privada Banfield S.A., Buenos Aires
  - 625-NOVAIN Neurociencias Group, Buenos Aires
  - 603-Fundación para el Estudio y Tratamiento de las Enfermedades Mentales - FETEM, Ciudad Autonoma Buenos Aires
  - 601-CENydET- Centro Neurobiologico y de Estres Traumatico-Biopsychomedical Research Group SRL, Ciudad Autonoma de Buenos Aire
  - 602-FunDamoS, Ciudad Autonoma de Buenos Aire
  - 622-Instituto Medico Damic Srl, Córdoba
  - 624-Centro Especializado en Neurociencias CEN, Córdoba
  - 626-Sanatorio Prof. Leon S. Morra S.A., Córdoba
  - 617-INSA Instituto de Neurociencias San Agustin S.A., La Plata
  - 623-Clinica Privada de Salud Mental Santa Teresa de Avila, La Plata
  - 607-Resolution Psicopharmacology Research Institute, Mendoza
- Bulgaria (22):
  - 454-Mental Health Centre 'Prof. Dr. Ivan Temkov', EOOD, Burgas
  - 533-State Psychiatric Hospital - Kardzhali, EOOD, Kardzhali
  - 532-MHAT "Dr. Hristo Stambolski", EOOD, Kazanlak
  - 569-State Psychiatric Hospital - Lovech, Lovech
  - 406-State Psychiatric Hospital - Pazardzhik AD, Pazardzhik
  - 535-UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - 586-Medical Center Mentalcare OOD, Plovdiv
  - 563-MC-Hipokrat-N E00D, Plovdiv
  - 403-University Multiprofile hospital for activated treatment Sveti Georgi, Clinic of psychiatry, Plovdiv
  - 592-Medical center Spectar - Plovdiv EOOD, Plovdiv
  - 570-Medical Centre "Sveti Naum", Sofia
  - 497-MHC - Sofia, EOOD, Sofia
  - 526-DCC "Sv. Vrach and Sv. Sv. Kuzma and Damyan", OOD, Sofia
  - 402-Military Medical Academy, Multiprofile Hospital for Actie Treatment - Sofia, Sofia
  - 405-UMHAT "Alexandrovska" EAD, Sofia
  - 568-Medical Center Hera EOOD, Sofia
  - 528-Medical Center Intermedica, OOD, Sofia
  - 404-MHAT-Targovishte, AD, Targovishte
  - 590-State Psychiatric Hospital - Tzarev Brod, Tsarev Brod
  - 498-DCC "Mladost M" - Varna, OOD, Varna
  - 455-Mental Health Center - Veliko Tarnovo EOOD, Veliko Tarnovo
  - 401-Mental Health Center-Vratsa EOOD, Vratsa
- Canada (3):
  - Chatham-Kent Clinical Trials Research Ctr, Chatham, Ontario
  - 351-McGill University Health Ctr Allan Memorial Int., Montreal, Quebec
  - 356-Chatham-Kent Clinical Trials Research Ctr, Chatham
- Croatia (5):
  - 536 - Clinic for psychiatry Vrapce, Zagreb
  - 537 - Clinic for psychiatry Vrapce, Zagreb
  - 550-Clinic for psychiatry Vrapce, Zagreb
  - 557 - Clinic for psychiatry Vrapce, Zagreb
  - 594-Klinika za psihijatriju Sveti Ivan, n/p Igor Filipčić or Marija Zelenika, Zagreb
- Czechia (6):
  - 512-NeuropsychiatrieHK s.r.o., Hradec Králové
  - 583-Narodni ustav dusevniho zdravi, Klecany
  - 519-A-SHINE s.r.o., Pilsen
  - 513-CLINTRIAL s.r.o., Prague
  - 499-MUDr. Tibor Miklos, Prague
  - 511-Psychiatrie Ricany s.r.o., Říčany
- Hungary (5):
  - 410-Dr. Máthé és Társa Bt., Kalocsa, Bács-Kiskun Megye
  - 411-ÓBudai Egészségűgyi Centrum Kft, Budapest, Pest County
  - 456-Semmelweis University Department of Psychiatry and Psychotherapy, Budapest, Pest County
  - 520-Nyiro Gyula Korhaz - Orszagos Pszichiatriai es Addiktologiai Intezet, Budapest
  - 440-PsychoTech Kft., Pécs
- Italy (2):
  - 566-Ospedale San Raffaele (San Raffaele Turro), Milan
  - 553-AO Città della Salute e della Scienza di Torino, Torino
- Lithuania (4):
  - 483-Romuvos klinika, UAB, Kaunas
  - 518-Kaunas City Outpatient Clinic, Public Institution, Kaunas
  - 484-Medical Center Puriena JSC, Šilutė
  - 517-Zirmunai Mental Health Center, Public Institution, Vilnius
- Poland (5):
  - 525-Podlaskie Centrum Psychogeriatrii, Bialystok
  - 502-Przychodnia Srodmiescie Sp. z o. o., Bydgoszcz
  - 579-Centrum Badan Klinicznych P.I. House Sp. z o.o., Gdansk
  - 501-Specjalistyczna Praktyka Lekarska Marek Domański, Lublin
  - 578-MSCZ im. Prof. J. Mazurkiewicza, Pruszków
- Russia (24):
  - 505-GUZ Lipetsk Regional psychoneurological Hospital #1, Plekhanovo, Lipetsk Oblast
  - 417-State Budget Healthcare Institution of Stavropol Region (Regional Specialized Psychiatric Hospital #2), Tonnel’nyy, Stavropol Kray
  - 418-State Budget Healthcare Institution of Arkhangelsk Region "Arkhangelsk Clinical Psychiatric Hospital", Arkhangelsk
  - 459-Federal State Budgetary Research Institution "Mental Health Science Center", Moscow
  - 573-SBIH of Moscow "Psychiatric Clinical Hospital # 4 n.a. P.B. Gannushkin" Short name: PCH N4 n.a. P.B.Gannushkin, Moscow
  - 581-SBIH of Moscow "Psych Clinical Hospital #1 N.A. Alekseev", Moscow
  - 419-State municipal healthcare Institution "Leningrad region psychoneurological center", Saint Petersburg
  - 415-Saint-Petersburg State Healthcare Institution "Saint Nicolas Wonderworker Psychiatric Hospital", Saint Petersburg
  - 571-St. Petersburg SHI "Psychoneurological Dispensary #10", Saint Petersburg
  - 451-V. M. Bekhterev National Research Medical Center For Psychiatry and Neurology, Saint Petersburg
  - 453-"Saint-Petersburg Scientific Research Psychoneurological Institute n.a. V.M. Bekhterev", Saint Petersburg
  - 465-"Saint-Petersburg Scientific Research Psychoneurological Institute N.A. V.M. Bekhterev", Saint Petersburg
  - 495-FSBI "National Medical Scientifi Center of Psychiatry and Neurology n.a. V.M. Bekhterev" MoH, Saint Petersburg
  - 464-Saint Petersburg State Budget Healthcare Institution "City Psychiatric Hospital No. 6 (Inpatient Department with Treatment Center)", Saint Petersburg
  - 443-Saint-Petersburg State Budget Healthcare Institution "Psychoneurological Center #5", Saint Petersburg
  - 444-SPHI "City Mental Hospital #3 n.a. I.I Skvortsov-Stepanov", Saint Petersburg
  - 452-Saint Petersburg State Public Institution of Healthcare "City Psychiatric Hospital #3 n.a.I.I. Skvortsov-Stepanov, Saint Petersburg
  - 496-SPHI "City Mental Hospital #3 n.a. I.I Skvortsov-Stepanov, Saint Petersburg
  - 458-State Budget Healthcare Institution "Samara Psychiatric Hospital", Saint Petersburg
  - 416-FSBEI HE "Smolensk State Medical University" of the MoH of the RF, Smolensk
  - 420-"Podderzhka" Research and Educational Center of Psychotherapy Limited Liability Company, Stavropol
  - 572-Klinika StoLet" Ltd., Tomsk
  - 466-OOO "Lion-Med", Voronezh
  - 422-State Budget Healthcare Institution of Yaroslavl Region "Yaroslavl Region Clinical Psychiatric Hospital", Yaroslavl
- Serbia (15):
  - 428-Clinical center of Serbia, Belgrade
  - 424-Institute of Mental health, Belgrade
  - 425-Clinical Hospital Center "Dr. Dragisa Misovic-Dedinje", Clinic of Psychiatry, Belgrade
  - 471-Clinic for Psychiatric Diseases "Dr Laza Lazarevic", Belgrade
  - 524-General Hospital Euromedik, Belgrade
  - 587-Institute of Mental Health, Belgrade
  - 584-Clinic for Psychiatry, Clinical Canter of Serbia, Belgrade
  - 472-Special Hospital for Psychiatric Diseases "Kovin", Kovin
  - 493-Special Neuropsychiatric Hospital Kovin, Kovin
  - 423-Clinical Center Kragujevac, Kragujevac
  - 429-Clinical Center Kragujevac, Clinic of Psychiatry, Kragujevac
  - 430-Psychiatric Clinic, Clinical Center Kragujevac, Kragujevac
  - 427-Clinical Center Nis, Clinic of Mental Health, Niš
  - 585-Special Hospital for Psychiatric Diseases "Gornja Toponica", Niš
  - 593-Specialized Hospital for Neuropsychiatric Diseases "Sveti Vracevi", Novi Kneževac
- Spain (8):
  - 476-FIDMAG Germanes Hospitalaries, Barcelona
  - 574-Hospital Clinic de Barcelona, Barcelona
  - 588-Institucion Hospitalaria Hestia Palau - Ensayos clinicos, Barcelona
  - 475-Hospital Gregorio Marañon, Madrid
  - 575-Hospital Universitario 12 de Octubre, Madrid
  - 494-CSM La Corredoria, Oviedo
  - 431-Centro de Salud Parquesol, 2ª planta - Servicio de Psiquiatria, Valladolid
  - 529-Hospital Provincial de Zamora, Zamora
- Ukraine (19):
  - 438-Communal Establishment "Odesa Regional Psychiatric Hospital #2", Odesa, Oblast
  - 462-Communal Establishment "I.I. Mechnykov Dnipropetrovsk Regional Clinical Hospital", Dnipro
  - 510-CI of Kyiv RC Regional Psychiatric-Narcological Medical Association, Depart #10 (male), Dept #2 (female), Hlevakha
  - 433-SI "Institute of Neurology, Psychiatry and Narcology of National Academy of Medical Sciences of Ukraine", Kharkiv
  - 434-State Institution "Institute of Neurology, Psychiatry and Narcology of NAMS of Ukraine", Department of Urgent Psychiatry and Narcology, Kharkiv
  - 582-SI Institute of Neurology,Psychiatry&Narcology of NAMSU, Kharkiv
  - 567-CIH Kharkiv Regional Clinical Psychiatric Hospital #3 Psychiatric Department of Primary Psychotic Episod Short Site name: CIH KRCPH #3 PD of PPE, Kharkiv
  - 461-Kherson Regional Psychiatric Hospital, Kherson
  - 507-Main Military Clinical Hospital of MDU, Kyiv
  - 447-Ukrainian Scientific Research Institute of Social and Forensic Psychiatry and Narcology of Ministry of Healthcare of Ukraine, Kyiv
  - Kyiv Regional Medical Incorporation Psychiatry Center of Novel Treatment and Rehabilitation of Psychotic Disorders, Department #29, Department #30, Kyiv
  - 460-Kyiv City Psychoneurological Hospital #3, General Psychiatry Department No. 2, Kyiv
  - 435-Kyiv Regional Medical Incorporation "Psychiatry". Center of Novel Treatment and Rehabilitation of Psychotic disorders, build 5, Department #30, Kyiv
  - 564-Regional Clinical Psychiatric Hospital, Nove
  - 509-CI Odesa Regional Medical Centre of Mental Health, Odesa
  - 508-CI Cherkasy Regional Psychiatric Hospital of ChRC Female Dept #11, Male Dept #12, Smila
  - 591-Municipal non-profit enterprise "Transcarpathian Regional Medical Center of Mental Health and Medicine of Addictions" of the Transcarpathian Regional Council, Department of psychiatry, Uzhhorod
  - Communal Establishment "Acad. O.I. Iushchenko Vinnytsia Regional Psychoneurologic Hospital", Vinnytsia
  - 432-Municipal Institution "Vinnytsya Regional Psychoneurological Hospital n.a. Acad. O.I. Yushchenko", Male Department No 14, Female Department No 15, Vinnytsya National Medical University n.a. M.I. Pyrogov, Dept of Psychiatry, Narcology and Psychothera, Vinnytsia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label extension study for patients from studies ACP-103-034, 038, and 064. Patients who had completed any of those studies and had not shown significant worsening of symptoms, or who may have benefited, or were expected to benefit from continued pimavanserin treatment based on the investigator's judgment were eligible.
Groups:
- Rollover From ACP-103-034; Rollover From ACP-103-038: Starting dose of 20 mg at week 1. The dose could be continued, decreased to 10 mg, or increased to 34 mg at investigator discretion through Week 52.
- Rollover From ACP-103-064: Pimavanserin dose of 34 mg throughout the study.
Period: Overall Study
Arm/Group | Rollover From ACP-103-034 | Rollover From ACP-103-038 | Rollover From ACP-103-064
Started | 323 | 325 | 347
Completed | 248 | 280 | 217
Not Completed | 75 | 45 | 130
Not completed — Study terminated by sponsor | 0 | 0 | 99
Not completed — Withdrawal by Subject | 37 | 14 | 9
Not completed — Not further specified | 6 | 11 | 10
Not completed — Adverse Event | 16 | 5 | 6
Not completed — Protocol Violation | 0 | 5 | 0
Not completed — Lack of Efficacy | 3 | 3 | 1
Not completed — Physician Decision | 2 | 2 | 0
Not completed — Noncompliance with study drug | 5 | 3 | 5
Not completed — Lost to Follow-up | 4 | 2 | 0
Not completed — Death | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Rollover From ACP-103-034 | Rollover From ACP-103-038 | Rollover From ACP-103-064 | Total
Number analyzed (Participants) | 323 | 325 | 347 | 995
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (9.30) | 37.8 (9.32) | 38.0 (9.47) | 37.7 (9.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 202 | 215 | 208 | 625
  Male | 121 | 110 | 139 | 370
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 25 | 13 | 0 | 38
  White | 295 | 309 | 346 | 950
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 1 | 4
Region of Enrollment [Number; unit: participants]
  North America | 45 | 29 | 0 | 74
  Europe | 278 | 296 | 284 | 858
  South America | 0 | 0 | 63 | 63

OUTCOME MEASURES:

1. Primary Outcome: Treatment Emergent Adverse Events
Description: Number of patients with treatment emergent adverse events
Time Frame: Treatment period (52 weeks) and follow-up period (30 days): planned total of 56 weeks. Since the study was prematurely terminated, the reporting period was shortened; AEs were assessed to the end of treatment, at a mean duration of 319 days (or 46 weeks).
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Groups:
- Rollover From ACP-103-064: Pimavanserin dose of 34 mg throughout the study (Week 26)
Arm/Group | Rollover From ACP-103-034 | Rollover From ACP-103-038 | Rollover From ACP-103-064
Number analyzed (Participants) | 323 | 325 | 347
Participants | 128 | 111 | 110

ADVERSE EVENTS:
Time Frame: Treatment period (52 weeks) and follow-up period (30 days): planned total of 56 weeks. Since the study was prematurely terminated, the reporting period was shortened; AEs were assessed to the end of treatment, at a mean duration of 319 days (or 46 weeks).
Description: This was an open-label extension study with assessment of safety/tolerability as primary objective. Inferential statistics was not planned. The study was terminated prematurely due to business reasons; mean follow-up duration of patients was shorter than specified in the protocol. Therefore, it was considered adequate to analyse pooled data, i.e. regardless of the trial from which patients originated or dose and dosing regimen patients used in this study.
Arm/Group | Rollover From ACP-103-034 | Rollover From ACP-103-038 | Rollover From ACP-103-064
All-Cause Mortality (participants affected / at risk) | 2/323 | 0/325 | 0/347
Serious Adverse Events (participants affected / at risk) | 13/323 | 4/325 | 4/347
Other Adverse Events (participants affected / at risk) | 21/323 | 30/325 | 19/347
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rollover From ACP-103-034 (N=323) | Rollover From ACP-103-038 (N=325) | Rollover From ACP-103-064 (N=347)
Dental cyst (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Drowning (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Tongue neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Schizophrenia (Psychiatric disorders) | 3 (3) | 1 (1) | 3 (3)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Psychiatric decompensation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rollover From ACP-103-034 (N=323) | Rollover From ACP-103-038 (N=325) | Rollover From ACP-103-064 (N=347)
Headache (Nervous system disorders) | 21 (23) | 30 (36) | 19 (24)

LIMITATIONS AND CAVEATS:
The study was terminated prematurely by the sponsor for business reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the study results, relative to their own patients, only after review, comment and approval by the sponsor. No publication of confidential information shall be made without the sponsor's prior written consent. At least 60 days prior to submitting a manuscript or prior to any public presentation, a copy of the manuscript or presentation will be provided to the Sponsor for review and comment. The sponsor has 60 days to review and comment.

DOCUMENTS (2):
  • Study Protocol (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT03121586/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-26): https://cdn.clinicaltrials.gov/large-docs/86/NCT03121586/SAP_001.pdf